CLINICAL TRIAL: NCT02681159
Title: Critical Incidents Related to Anesthesia and Intensive Care: A Prospective Study in a Tertiary Hospital
Brief Title: Critical Incidents Related to Anesthesia and Intensive Care: A Study in a Tertiary Hospital
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Subhi M. Alghanem, Professor of Anesthesia and Intensive Care, University of Jordan
Other Study IDs: 272/14a/tk
Record Dates: First submitted 2016-01-28; First posted 2016-02-12 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Critical Incident
Keywords: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
Critical incidents in anesthesia is one of the most valuable methods to assess the safety of anesthesia practice among different types of patients. Most of the studies in this regards are retrospective with many drawbacks and pitfalls like absence of information in the records of the patients.

In the investigators' study, the investigators will follow the critical incidents among patients who underwent surgery under anesthesia whether regional or general over the next two years from 2016 to 2018, by examining the patients records from the hospital database and recording the events that occur to the patients.

DETAILED DESCRIPTION:
Over the forthcoming two years, the investigators will study in details critical incidences that may occur to patients in the perioperative period like; acute hypoxic event, acute major hemorrhage, acute airway obstruction and others that may endanger the life or one of the patient organs and whether the patient survive the acute event or die.

These critical incidences will be collected and all information about it will be known in order to be studied and to know were was the defect and eventually to improve the safety of practice of anesthesia and surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo anesthesia and surgery
* patients who are exposed to a critical incidence

Exclusion Criteria:

* patients who undergo anesthesia and surgery and do not expose to critical incidents.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who undergo anesthesia and surgery and be exposed to a critical incidence.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
number of anesthetized patients who have perioperative critical incidence. | 14 days
  Critical incidence will include:
  Aspiration , Laryngospasm , Hypoxemia, Hypoventilation , Hypertension , Hypotension, Myocardial ischemia / infarction, Cardiac arrhythmia, Acute cardiac decompensation , Dental lesion , Nerve / skin / cornea lesion , Lesion through needle puncture , Hypothermia , Conversion of regional anesthesia / inadequate block, Urinary retention , Inadequate postoperative analgesia , Postoperative agitation ,) Awareness , Allergic reaction, Transfusion / mediation error, Miscellaneous.

CONTACTS AND LOCATIONS:
Overall Officials: Subhi M Alghanem, FFARCS, Study Chair — University of Jordan
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munting KE, van Zaane B, Schouten AN, van Wolfswinkel L, de Graaff JC. Reporting critical incidents in a tertiary hospital: a historical cohort study of 110,310 procedures. Can J Anaesth. 2015 Dec;62(12):1248-58. doi: 10.1007/s12630-015-0492-y. Epub 2015 Sep 25. PMID 26407581